CLINICAL TRIAL: NCT02674867
Title: ANRS EP59 CLEAC : Physiopathological Study of Immunovirological Evolution of Perinatally HIV-1 Infected Children Depending on Early (Before 6 Months) or Late (After 2 Years) Antiretroviral Therapy Introduction.
Brief Title: CLEAC (Comparison of Late Versus Early Antiretroviral Therapy in HIV-infected Children)
Acronym: CLEAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS EP 59 CLEAC
Record Dates: First submitted 2016-01-13; First posted 2016-02-05 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early treatment group (Experimental): Vertically-HIV-1-infected children, between 5 and 17-year-of-age, who started cART before 6 months-of-age ("early treatment" group) with an initial virologic success (HIV-1 RNA <400 copies / mL reached no later than 24 months after the start of cART), whatever the later evolution of the viremia.
  Interventions: Other: Blood draw
- Late treatment group (Other): Vertically-HIV-1-infected children, between 5 and 17-year-of-age, who started cART after 24 months-of-age ("late treatment" group) with an initial virologic success (HIV-1 RNA <400 copies / mL reached no later than 24 months after the start of cART), whatever the later evolution of the viremia.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw

SUMMARY:
The study aims to define and compare the immunological characteristics (lymphocyte subpopulations, specific immunity against HIV, lymphocyte activation, inflammatory parameters) and the virological characteristics (study of viral reservoir) between 2 groups of vertically-HIV-1-infected children, between 5 and 17-year-of-age, who started cART before 6 months-of-age ("early treatment" group) or after 24 months-of-age ("late treatment" group) with an initial virologic success (HIV-1 RNA <400 copies / mL reached no later than 24 months after the start of cART), whatever the later evolution of the viremia.

Moreover, the viral reservoir will be deeply characterized in 10 children (5 patients in each group) with sustained control of the HIV-1 viremia under cART (≥ 90% of HIV-1 RNA measures <400 copies /mL): quantification of the reservoir in the lymphocyte subpopulations and study of the inductibility of the viral reservoir.

DETAILED DESCRIPTION:
This is a cross-sectional study, multicenter, without direct benefit, among vertically HIV-1 infected children, aged 5 to 17 years, followed in centers participating in the ANRS CO10 EPF cohort located in Ile-de-France. Eligible children are not necessarily included in the cohort. The sample will consist of two age groups of equal size (5-12 years and 13-17 years).

Patient recruitment will be conducted in the centers of the ANRS CO10 EPF cohort located in Ile de France (Paris area). 80 children will be included, previously included or not in the ANRS CO10 EPF cohort. Our investigations will involve two blood samples, taken during two successive visits of the children in the hospitals where they are usually followed. Finally, a third blood sample will be taken during a third visit only for the 10 children participating in the substudy of the viral reservoir. All medical data since birth will be prospectively collected for children included in the ANRS CO10 EPF cohort, and retrospectively collected in the other cases.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 17 years old
* Vertically HIV-1 infected, not HIV-2 co-infected
* Diagnosed < 13 years old
* Usually followed in a center participating in the ANRS CO10 EPF cohort located in Ile de France
* Have received cART treatment:

  * started later than 6 months-of-age ("early treatment" group) or after 24 months-of-age ("late treatment" group)
  * with an initial virologic success (HIV-1 RNA <400 copies / mL reached no later than 24 months after the start of cART),
* Affiliated person or beneficiary of a social security system (Article L1121-11 of the Code of Public Health) (medical aid of state or AME is not a social security system)
* Participant agreement if in age to give an opinion
* Free, informed and written consent, signed by at least one parent and the investigator

Exclusion Criteria:

* < 5 years old or ≥ 18 years old at first sample for the study
* Obviously HIV-1 infected after the perinatal period
* HIV-2 co-infected
* Diagnosed ≥ 13 years old
* Started cART treatment between 7 and 23 months
* No HIV-1 RNA <400 copies / mL within 24 months after initiation of treatment (considered as a failure of the first line therapy)
* Not affiliated to the French social security, or beneficiary of a social security system
* Refusal to participation of parent(s) (or the holders(s) of parental authority)
* Refusal to participation if in age to give an opinion.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Immune status | Baseline
  The immune status will be defined by T lymphocyte subpopulations
Virological status | Baseline
  Peripheral blood HIV DNA levels
Immune status | 6 months after baseline
  The immune status will be defined by inflammatory parameters : cytokines and chemokines
Immune status | Baseline
  The immune status will be defined by HIV-specific T cell response
Immune status | Baseline
  The immune status will be defined by lymphocyte activation (HLA-DR)

SECONDARY OUTCOMES:
Comparison of immune and virological statuses of early and late treatment groups | Baseline
  Two groups of vertically-HIV-1-infected children, between 5 and 18-year-of-age, will be compared: the "early treatment" group that comprises children who started HAART before 6 months-of-age, and the late treatment" group those who started HAART after 24 months-of-age.
Viral reservoir : lymphocyte subpopulation | One year after baseline
  Total HIV- DNA will be quantified by ultrasensitive PCR in CD4 T cell subsets sorted according their differenciation status for 10 children (5 patients in each group) with sustained control of the HIV-1 viremia under HAART ( ≥ 90% of HIV-1 RNA measures <400 copies / ml).
Viral reservoir : inductibility | One year after baseline
  Inductibility of the viral reservoir will be quantified by ultrasensitive HIV-RNA RT- PCR in supernatants after coculture of CD4 T cells.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Hôpital Jean Verdier, Bondy
  - Hôpital Louis Mourier, Colombes
  - Centre Hospitalier Intercommunal, Créteil
  - Centre hospitalier Francilien Sud, Évry
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Groupe hospitalier Cochin Port Royal, Paris
  - Groupe Hospitalier Necker, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Trousseau, Paris
  - Centre Hospitalier Général- Hôpital Delafontaine, Saint-Denis
  - Centre Hospitalier Général, Villeneuve-Saint-Georges

REFERENCES:
- [Derived] Frange P, Montange T, Le Chenadec J, Batalie D, Fert I, Dollfus C, Faye A, Blanche S, Chace A, Fourcade C, Hau I, Levine M, Mahlaoui N, Marcou V, Tabone MD, Veber F, Hoctin A, Wack T, Avettand-Fenoel V, Warszawski J, Buseyne F. Impact of Early Versus Late Antiretroviral Treatment Initiation on Naive T Lymphocytes in HIV-1-Infected Children and Adolescents - The-ANRS-EP59-CLEAC Study. Front Immunol. 2021 Apr 22;12:662894. doi: 10.3389/fimmu.2021.662894. eCollection 2021. PMID 33968064